CLINICAL TRIAL: NCT04505215
Title: Comparison of the Effect of Mulligan and Muscle Energy Techniques on Pain, Grip Strength and Functionality in Individuals With Lateral Epicondylitis
Brief Title: Comparison of Mulligan Technique and Muscle Energy Technique in Lateral Epicondylitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KaratayUS
Record Dates: First submitted 2020-07-23; First posted 2020-08-10 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2020-08

CONDITIONS: Tennis Elbow
Keywords: Tennis Elbow; Exercise; Musculoskeletal Manipulations
MeSH Terms: conditions — Tennis Elbow; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mulligan Technique (Experimental): In addition to the exercises applied to the participants in the control group, the participants in this group used Mobilization with movement, which was performed with the principle of painless movement 3 times a week for a total of 12 times a week for 4 weeks. Mobilization with movement has been performed by a certified physiotherapist who has been practicing this technique for 10 years.
  Interventions: Other: Mulligan Technique
- Muscle Energy Technique (Experimental): In addition to the exercises applied to the participants in the control group, the Janda method (Post Isometric Relaxation Technique) from Muscle Energy Technique (3 times a week) was used 3 times a week for 4 weeks.
  Interventions: Other: Muscle Energy Technique
- Only Exercise (Control) (Active Comparator): Stretching and strengthening exercises for the forearm extensors were shown to the participants in the control group for 4 weeks every day of the week.
  Interventions: Other: Only Exercise (Control)

INTERVENTIONS:
Other: Mulligan Technique — First, the painless application angle was determined for each patient. The lateral condyle of the humerus was fixed by the web range of the physiotherapist. The elbow joint was glided until the elbow joint and the hand tightening position were not able to cause pain.
  The patients were asked to repeat the motion of the elbow joint and the ball squeezing motion given to their hands 10 times without pain. For pain control, the same procedure was performed with three sets, each containing 10 repetitions of the exercise. The interval between sets was 15 to 20 seconds, and the interval between repetitions within each set was 30 seconds.
  Arms: Mulligan Technique
Other: Muscle Energy Technique — Firstly, 5-7 sec opposite isometric muscle contraction was requested from the patient in the barrier by passively stretching by the physiotherapist until the barrier of the related muscle or dysfunctional joint. After a short rest period of 2-3 seconds, the physiotherapist continued to stretch passively until the second barrier. The application continued until the tension of the muscle or dysfunction of the joint disappeared.
  Arms: Muscle Energy Technique
Other: Only Exercise (Control) — Eccentric training for the extensor Carpi Radialis Brevis (ECRB) muscle, the most affected wrist extensor tendon, and static stretching exercise for the EKRB muscle were given as home exercise program. The best stretching position for the EKRB tendon is provided when the elbow joint is in extension, forearm pronation, when the wrist is flexed with ulnar deviation (Mills maneuver). Each exercise was taught to patients in 10 repetitions and 10 seconds, and one day of the week, participants in the control group performed their exercises under the supervision of a physiotherapist.
  Arms: Only Exercise (Control)

SUMMARY:
In this study, the effects of mulligan and muscle energy techniques on pain, grip strength and functionality will be investigated in a randomized controlled manner in individuals with lateral epicondylitis. Various treatments have been tried in patients with lateral epicondylitis whose daily activities are restricted in order to reduce pain and increase functions. Among them, conservative and physical therapy agents have an important place. There are many studies in the literature evaluating the effects of mobilization in LE treatment. However, there are no definitive data on the long-term efficacy and benefits of all these treatment methods. Mulligan and muscle energy techniques can be used in lateral epicondylitis due to many positive reasons such as being effective in a short time, giving fast results, high success rate, risk-free and painless in the case of specialists. Thanks to the findings obtained from our study, it is aimed to contribute to the literature with objective, evidence-based results in this field.

DETAILED DESCRIPTION:
Lateral epicondylitis (LE); It is one of the most common lesions of the upper limb, originating from the wrist and wrist extensor muscles, characterized by pain in the lateral epicondyle and extensor muscle surface of the forearm. LE was first described by Runge in 1873 and was named tennis elbow by Morris in 1882. It is thought that the cause of LE is caused by repetitive stresses, direct traumas, repetitive contractions, degeneration, micro tears, immature repair and tendinosis at the adhesion of the extensor carpi radialis brevis and extensor digitorum communis muscles. It is mostly seen in 4-6 decades. More dominant upper limb is affected. Its annual incidence has been determined between 1-3%. It has been shown that it can cause a significant loss of labor due to pain in patients.

The Mulligan Concept is a new approach in Manual Therapy. It was started to be developed by New Zealand physiotherapist Brian Mulligan in the 1980s, and its popularity and awareness has increased in the last 10 years. The concept-specific techniques called NAGS, SNAGS and MWMs are applied safely and effectively in musculoskeletal-nervous system diseases. The concept is suitable for biomechanics, arthrokinematic kinesiological principles, which are the common knowledge of the known Manual Therapy approaches, and techniques and application principles are important with other approaches. show differences.

Manual therapy and forearm extensor muscle strengthening are used together with MWM (mobilization with movement) technique. MWM eliminates elbow pain by reducing abnormal facilitations and creates some tactile and compressive stimuli in soft tissue. Afferent nerve activity results in these tactile and compressive stimuli inhibiting spinal cord neurons. Force is applied at long load at low load. Increases the harmony and mobility of connective tissue layers.

Mulligan concept; It can be defined as a combination of passive mobilization concepts such as Kaltenborn, Maitland Cyriax, and active methods such as Pilates, PNF and Kinetic Control. The distinctive feature of this approach is that, when the right case is chosen, the pain can be achieved, functional gains can be achieved in a very short time and in the long term.

Postisometric reconstruction: muscle energy technique (MET) is a manual therapy that uses muscle's own energy in the form of mild isometric contractions to relax and lengthen muscles through autogenic or mutual inhibition. Compared to static stretching, a passive technique in which the therapist does all the work, MET is an active technique in which the patient is also an active participant. BAT is based on the concepts of Autogenic Inhibition and Mutual Inhibition. If a maximum contraction of the muscle is followed by the stretching of the same muscle, Autogenic Inhibition is known as MET, and if the opposite muscle following a maximum contraction of the muscle is stretched, it is known as Mutual Inhibition MET.

The manipulative treatment acts directly on the joint structures and creates a nociceptive afferent stimulation by providing physiological effect on the central nervous system. Such findings emphasize the appropriateness of the local movements of mobilization. Such a mechanism may include intranoral circulation, axoplasmic flow, or neural connective tissue viscoelasticity. However, an increasing number of studies have shown that passive joint movements can activate many areas.

Exercise programs are the most common physiotherapy treatments for LE. There are many studies examining the effects of exercise programs in LE. Stretching and strengthening exercises are at the core of the exercise program. Because the tendon should not only be strengthened, it should be flexible. Home exercises should usually be done once or twice a day.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosing lateral epicondylitis
* Age between 30 and 60 years
* Willingness to comply with treatment and follow-up assessments

Exclusion Criteria:

* Treatment of elbow complaints with surgical intervention
* Physiotherapy or CSIs in the past 6 months
* Duration of <3 months
* Severe neck or shoulder problems likely to cause or maintain the elbow complaints
* Posterior interosseous nerve compression
* Congenital or acquired deformities of the elbow
* Systemic musculoskeletal or neurologic disorders

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2020-08-14 (Actual); Primary Completion 2020-11-07 (Actual); Study Completion 2020-11-14 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Hand Grip Strenght at 6 weeks | Baseline and 4 weeks
  The maximum grip force measurements of the patients were made with "Baseline Hydraulic Hand Dynamometer". The patient's measurements were carried out in two positions. While the patient was in a sitting position, measurements were made in shoulder adduction, elbow 90˚ flexion, forearm in neutral position, wrist in 0-30˚ extension and 0-15˚ in ulnar deviation position. While the patient was standing, measurement was performed with shoulder adduction, elbow extension, forearm in neutral position. For maximum grip, patients should be able to hold the dynamometer for a maximum of 3 seconds. it was said to tighten with all its might. Measurements were repeated 3 times at 30-second intervals on the affected limb, and the measurements were averaged. Values are noted in kilograms (kg) - force
Change from baseline in Pain Score at 6 weeks | Baseline and 4 weeks
  Visual Analogue Scale was used to determine the severity of rest, activity and night pain in patients with lateral epicondylitis. Patients were asked to mark their pain levels on a 10 cm scale before starting treatment and after 4 weeks of treatment. The value "0" means that there is no pain, and the value "10" means unbearable pain. The marked points are measured and recorded in centimeters

SECONDARY OUTCOMES:
Change from baseline in Functionality at 6 weeks | Baseline and 4 weeks
  Patient-rated Forearm Evaluation Questionnaire Overend et al. It was designed to evaluate treatment specifically for patients with lateral epicondylitis. Afterwards, it was rearranged by the same working group and named as Patient-rated Forearm Evaluation Questionnaire. The survey consists of 15 questions that question patients' difficulties and pain in the past week. Pain level (5 questions), elbow-related functions (6 questions, special activities, 4 questions daily activities) are evaluated in the first section. The total score ranges from 0 to 100, and high scores indicate increased pain and loss of functionality. In 2010, Altan et al. Turkish version was created by, Patient-rated Forearm Evaluation Questionnaire was found valid and reliable. Turkish version of the questionnaire was used in our study.

CONTACTS AND LOCATIONS:
Overall Officials: Bayram Sönmez ÜNÜVAR, Principal Investigator — KTO Karatay University
Locations (1):
- KTO Karatay University, Konya, Turkey (Türkiye)